CLINICAL TRIAL: NCT03769337
Title: Identification of New Biological Marker for Diagnosis of Periprosthetic Infections
Brief Title: New Markers for Diagnosis of Prosthetic Infections
Acronym: Perimarkers
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: I.R.C.C.S Ospedale Galeazzi-Sant'Ambrogio (Other)
Responsible Party: Sponsor
Other Study IDs: Perimarkers
Record Dates: First submitted 2018-12-06; First posted 2018-12-07 (Actual); Last update posted 2018-12-24 (Actual); Status verified 2018-11

CONDITIONS: Prosthetic Joint Infections
Keywords: serum markers of infections

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Serum
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Infected: Serum biomarkers in patients with diagnosis of prosthetic joint infection
  Interventions: Diagnostic Test: serum biomarkers
- Not Infected: Serum biomarkers in patients with implant failure not caused by infection
  Interventions: Diagnostic Test: serum biomarkers

INTERVENTIONS:
Diagnostic Test: serum biomarkers — Measurement of Serum concentrations of IL-6, TREM-1, CCL2, MMP-9, OPN, IL-1RA, GP-130, C5a, sRAGE, urokinase and presepsin before revision surgery and after 2 and 7 days after surgery

SUMMARY:
Implant infections are among the most dramatic complications in orthopaedic surgery with heavy impact on life quality and health system. Their diagnosis is still challenging since, till now, none othe proposed markers has shown a sensitivity and a specificity of100%. Therefore, efforts in identification of new markers of infections are required. This study aims to evaluate the applicability of Interleukin (IL)-6, Triggering receptor expressed on myeloid cells (TREM-1), CC chemokine ligand 2 (CCL2), matrix metalloproteinases (MMP-9), osteopontin (OPN), IL-1 receptor antagonist (IL1-RA), IL-6 receptor beta (GP130), C5a, receptor for advanced glycation end products (sRAGE), urokinases and presepsin as serum markers of prosthetic joint infection.

At this purpose, serum from 65 patients with infected implant and from 65 with aseptic failure of their prosthesis will be collected before surgery and after 2 and 7 days from revision.

DETAILED DESCRIPTION:
Management of prosthetic joint infections involves long antibiotic therapy and, in most cases, additional revision surgery with worsening of life quality for patients and high costs for health system. Prosthetic joint infections occur at a rate of 1-2% but their incidence grows up to 15-20% after the first revision surgery. Gram positive cocci, particularly staphylococci, are the main pathogens responsible for these infections. Diagnostic workflow is rather complicated, since a gold standard assay characterized by high sensitivity and specificity has not been recognized. Consequently, the diagnosis is based on fulfillment of a series of major and minor criteria derived from biochemical, hematological, microbiological, histological analyses combined with clinical and radiological observations. Therefore, it is evident that there is an urgent need to find early markers of infection, characterized by high sensitivity and specificity able to differentiate between aseptic failure and prosthetic joint infections caused by both high and low virulent microorganisms.

In the recent years, presepsin has been described as a marker for sepsis also able to discriminate sepsis severity. Presepsin is a fragment of soluble receptor CD14 which is released from monocyte surface during inflammation. The new inflammatory marker TREM-1 links the activity of presepsin to other actors of inflammation process like Toll Like Receptors, monocytes, inflammatory cytokines like IL-1 and IL-6, the chemokine CCL2. Presepsin activity is also related to suPAR an inflammatory marker, we have recently shown to be associated with prosthetic joint infections. Another potential marker of infection is osteopontin (OPN), a multifunctional protein with pro-inflammatory properties, which correlates with mortality and is associated to suPAR in inflammatory response. Similarly, receptor CD163, highly expressed by macrophages during inflammation has been proposed as a promising serum marker of inflammation. Equally important in inflammatory process is the role played by neutrophils, which represent the first line of defense against infection, being able to kill bacteria by producing oxygen reactive species (ROS). Recently ROS have been correlated with serum Advanced Glycation End Products(AGEs) that are increased by oxidative stress. AGEs are able to interact with their receptor RAGE, which exists in its soluble forms in plasma. For this reason, RAGE might be used as serum biomarker to diagnose infection and related oxidative stress. Despite the amount of scientific papers on the role of the above mentioned molecules, a panel combining them for diagnosis of prosthetic joint infections is not yet available.

Aim of the study will be to evaluate new biological markers of prosthetic joint infection in order to improve diagnostic workflow to support and integrate data from microbiological, hematological and clinical examination.

At this purpose, differences in serum concentrations of IL-6, TREM-1, CCL2, MMP-9, OPN, IL-1RA, GP-130, C5a, sRAGE, urokinases and presepsin between infected and not infected patients will be evaluated by measuring sensitivity, specificity, positive and negative predictive values, likelihood ratio for each parameter. Moreover, concentration of each biomarker will be correlated with markers routinely used for diagnosis of these infections.

A total of 130 patients will be enrolled in the study: 65 patients with diagnosis of aseptic failure, and 65 diagnosed with infection of prosthetic implant.

All of them will sign an informed consent before enrollment. An aliquot of serum sent to the Laboratory for pre- and post-operative (2 and 7 days after surgery) routine analyses will be stored at -20°C.

Serum concentrations of IL-6, TREM-1, CCL2, MMP-9, OPN, IL-1RA, GP-130, C5a, sRAGE, urokinase and presepsin will be determined by means of commercially available ELISA assays.

Data regarding preoperative Erythrocyte Sedimentation Rate (ESR) and C-reactive protein (CRP), Synovial fluid analysis (if available, both pre and intra operative), and microbiological culture (implant and periprosthetic tissues) will be also collected.

ELIGIBILITY:
Inclusion Criteria:

* Patients with diagnosis of septic or aseptic failure of prosthetic implant
* Informed consent signed

Exclusion Criteria:

* Patients undergoing revision surgery for failure not due to the above mentioned causes
* Known auto immune diseases or other conditions which might alter inflammatory response

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with failure of prosthetic implant
Sampling Method: Non-Probability Sample
Enrollment: 130 (Estimated)
Dates: Start 2018-09-01 (Actual); Primary Completion 2020-08-31 (Estimated); Study Completion 2020-09-30 (Estimated)

PRIMARY OUTCOMES:
Statistically significant differences in serum concentrations of IL-6 between infected and not-infected patients | within 1 year after collection of all samples
  Serum concentrations of IL-6 will be compared before surgery and at 2 and 7 days after implant revision.
Statistically significant differences in serum concentrations of TREM-1 between infected and not-infected patients | within 1 year after collection of all samples
  Serum concentrations of TREM-1 in infected and not-infected patients will be compared before surgery and at 2 and 7 days after implant revision.
Statistically significant differences in serum concentrations of CCL-2 between infected and not-infected patients | within 1 year after collection of all samples
  Serum concentrations of CCL2 in infected and not-infected patients will be compared before surgery and at 2 and 7 days after implant revision.
Statistically significant differences in serum concentrations of MMP-9 between infected and not-infected patients | within 1 year after collection of all samples
  Serum concentrations of MMP-9 in infected and not-infected patients will be compared before surgery and at 2 and 7 days after implant revision.
Statistically significant differences in serum concentrations of OPN between infected and not-infected patients | within 1 year after collection of all samples
  Serum concentrations of OPN in infected and not-infected patients will be compared before surgery and at 2 and 7 days after implant revision.
Statistically significant differences in serum concentrations of IL-1RA, between infected and not-infected patients | within 1 year after collection of all samples
  Serum concentrations of IL-1RA in infected and not-infected patients will be compared before surgery and at 2 and 7 days after implant revision.
Statistically significant differences in serum concentrations of GP-130 between infected and not-infected patients | within 1 year after collection of all samples
  Serum concentrations of GP-130 in infected and not-infected patients will be compared before surgery and at 2 and 7 days after implant revision.
Statistically significant differences in serum concentrations of C5a between infected and not-infected patients | within 1 year after collection of all samples
  Serum concentrations of C5a in infected and not-infected patients will be compared before surgery and at 2 and 7 days after implant revision.
Statistically significant differences in serum concentrations of sRAGE between infected and not-infected patients | within 1 year after collection of all samples
  Serum concentrations of sRAGE in infected and not-infected patients will be compared before surgery and at 2 and 7 days after implant revision.
Statistically significant differences in serum concentrations of urokinase between infected and not-infected patients | within 1 year after collection of all samples
  Serum concentrations of urokinase in infected and not-infected patients will be compared before surgery and at 2 and 7 days after implant revision.
Statistically significant differences in serum concentrations of presepsin between infected and not-infected patients | within 1 year after collection of all samples
  Serum concentrations of presepsin in infected and not-infected patients will be compared before surgery and at 2 and 7 days after implant revision.

CONTACTS AND LOCATIONS:
Overall Officials: Elena De Vecchi, MSc, Principal Investigator — IRCCS Istituto Ortopedico Galeazzi
Locations (1):
- IRCCS Istituto Ortopedico Galeazzi, Milan, MI, Italy

IPD SHARING:
Plan to Share IPD: Yes
De-identified participants data for all primary outcome measures will be made available
Supporting Information: Study Protocol, SAP
Time Frame: Data will be made available within 1 year after completion of the study
Access Criteria: Data access request will be sent to the facility